CLINICAL TRIAL: NCT00534833
Title: Immunogenicity Study of the Antibody Persistence and Booster Effect of DTaP-Hep B-PRP-T Combined Vaccine or Tritanrix HepB/Hib™ at 15 to 18 Months of Age Following a Primary Series at 6, 10 and 14 Weeks of Age in Healthy Filipino Infants
Brief Title: Immunogenicity Study of Antibody Persistence and Booster Effect of DTaP-HB-PRP~T Combined Vaccine or Tritanrix-HepB/Hib™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AL205
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-09

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Haemophilus Influenzae Type b
Keywords: Diphtheria; Tetanus; Pertussis; Hepatitis B Hansenula (HB); Haemophilus influenzae type b
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Haemophilus Infections | interventions — diphtheria-tetanus-acellular pertussis-Hib-hepatitis B vaccine; Poliovirus Vaccine, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): DTaP-Hep B-PRP-T + OPV vaccine group
  Interventions: Biological: DTaP-HB-PRP~T vaccine; Biological: Oral Polio Vaccine
- Group 2 (Active Comparator): Tritanrix-HepB/Hib™ + OPV vaccine group
  Interventions: Biological: Tritanrix-HepB/Hib™; Biological: Oral Polio Vaccine

INTERVENTIONS:
Biological: DTaP-HB-PRP~T vaccine — 0.5 mL, Intramuscular
  Arms: Group 1
Biological: Tritanrix-HepB/Hib™ — 0.5 mL, Intramuscular
  Arms: Group 2
Biological: Oral Polio Vaccine — 0.5 mL, Oral

SUMMARY:
The present trial is a follow-up of AL203 study (NCT00343889).

Primary Objectives:

To describe the antibody persistence at 15 to 18 months of age and the booster effect of a dose of DTaP-HB-PRP~T or Tritanrix-HepB/Hib™ (given concomitantly with Oral Polio Vaccine [OPV]).

Secondary Objective:

To describe the safety profile of a booster dose of DTaP-HB-PRP~T or Tritanrix-HepB/Hib™ when administered concomitantly with OPV in each vaccine group.

DETAILED DESCRIPTION:
Study participants will receive a booster vaccination of DTaP-HB-PRP~T or Tritanrix-HepB/Hib™ either concomitantly with Oral Polio Vaccine (OPV) following the completion of a three dose primary series with DTaP-Hep B-PRP-T combined vaccine or Tritanrix HepB/Hib™, both given concomitantly with OPV. Participants will receive a booster dose of the vaccine they had received in the primary series, and a concomitant dose of OPV Study AL203 (NCT00343889).

ELIGIBILITY:
Inclusion Criteria:

* Toddler aged 15 to 18 months of age on the day of inclusion (range: 456 days to 578 days of age inclusive)
* Participated in the AL203 study and completed the three-dose primary series with either DTaP-HB-PRP~T or Tritanrix-HepB/Hib™, and OPV, at 6, 10 and 14 weeks of age
* Informed consent form signed by one parent or legal representative if appropriate (independent witness mandatory if parent is illiterate)
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term (for more than 2 weeks) systemic corticosteroid therapy within the preceding 3 months
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Blood or blood-derived products received in the last 3 months
* Any vaccination in the 4 weeks preceding the trial vaccination
* Vaccination planned in the 4 weeks following the trial vaccination
* Febrile (temperature ≥ 38.0°C) or acute illness on the day of inclusion
* History of documented diphtheria, tetanus, pertussis, Haemophilus influenzae type b, hepatitis B or poliomyelitis infection(s) (confirmed either clinically, serologically, or microbiologically)
* Vaccination with a vaccine containing diphtheria, tetanus, pertussis, Haemophilus influenzae type b, hepatitis B, or poliovirus 3 types antigen since the end of the primary series
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular (IM) vaccination
* Serious adverse event related to any vaccination in the AL203 study.

Ages: 15 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Philippines (2):
  - Manila
  - Quezon City

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized and enrolled from 21 September 2007 to 03 December 2007 in 2 clinical centers in the Philippines.
Pre-assignment Details: A total of 362 participants who met the inclusion but not the exclusion criteria were enrolled and vaccinated.
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received a booster dose of DTaP-Hep B-PRP~T concomitantly with OPV at age 15 to 18 months following a three dose primary series of DTaP-Hep B-PRP~T combined vaccine given concomitantly with OPV at 6, 10, and 14 weeks of age in the AL203 study.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received a booster dose of Tritanrix-Hep B/ Hib™ concomitantly with OPV at age 15 to 18 months following a three dose primary series of Tritanrix-Hep B/ Hib™ combined vaccine given concomitantly with OPV at 6, 10, and 14 weeks of age in the AL203 study.
Period: Overall Study
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Started | 182 | 180
Completed | 182 | 180
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received a booster dose of DTaP-Hep B-PRP-T concomitantly with Oral Polio Vaccine (OPV) at age 15 to 18 months following a three dose primary series of DTaP-Hep B-PRP-T combined vaccine given concomitantly with OPV at 6, 10, and 14 weeks of age in the AL203 study.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received a booster dose of Tritanrix-Hep B/ Hib™ concomitantly with Oral Polio Vaccine (OPV) at age 15 to 18 months following a three dose primary series of Tritanrix-Hep B/ Hib™ combined vaccine given concomitantly with OPV at 6, 10, and 14 weeks of age in the AL203 study.
- Total: Total of all reporting groups
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV | Total
Number analyzed (Participants) | 182 | 180 | 362
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 182 | 180 | 362
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Months] | 15.9 (0.946) | 15.9 (0.942) | 15.9 (0.945)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 88 | 185
  Male | 85 | 92 | 177
Region of Enrollment [Number; unit: Participants]
  Philippines | 182 | 180 | 362

OUTCOME MEASURES:

1. Primary Outcome: Summary of Antibody Persistence and Immunogenicity Booster Response in Participants Who Were Vaccinated With Either DTaP-Hep B-PRP~T Concomitantly With Oral Polio Vaccine (OPV) or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Immunogenicity was assessed by means of radioimmunoassay (RIA) for anti-Hepatitis B (Hep Bs) and anti-polyribosyl ribitol phosphate (PRP) antibodies, enzyme immunoassay (EIA) for anti-Tetanus, and serum neutralization for anti-Diphtheria.
  Booster responses defined as titers ≥ 10 mIU/mL for anti-Hep Bs; ≥ 0.15 μg/mL for anti-PRP; ≥ 0.01 IU/mL for anti-Tetanus and anti-Diphtheria at Day 28 after the third vaccination; Pertussis Toxoid (PT) and Filamentous Hemagglutinin (FHA) 4-fold increase, and individual titers ratio.
Time Frame: 28 Days post-vaccination
Population: Antibody persistence and immunogenicity booster responses were assessed in a subset of participants available for the endpoint, the per-protocol population.
Measure: Number; unit: Participants
Groups:
- Group 1: DTaP-Hep B-PRP~T + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine following a 3-dose primary series of DTaP-Hep B-PRP~T combined vaccine concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL203.
- Group 2: Tritanrix-Hep B/ Hib™ + OPV: Participants received a booster dose of the DTaP-Hep B-PRP~T Combined vaccine following a 3-dose primary series of Tritanrix-Hep B/ Hib™ concomitantly with OPV at 6, 10, and 14 weeks of age in Study AL203
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 98 | 98
Participants
  Anti-Hep B, Pre-booster (N = 98, 98) | 36 | 58
  Anti-Hep B, Post-booster (N = 98, 98) | 81 | 94
  Anti-PRP, Pre-booster (N = 98, 98) | 82 | 97
  Anti-PRP, Post-booster (N = 98, 98) | 97 | 98
  Anti-Diphtheria, Pre-booster (N = 98, 98) | 67 | 59
  Anti-Diphtheria, Post-booster (N = 98, 98) | 97 | 97
  Anti-Tetanus, Pre-booster (N = 98, 97) | 98 | 97
  Anti-Tetanus, Post-booster (N = 98, 98) | 98 | 98
  Anti-Pertussis, 4-Fold Increase (N = 96, 92) | 94 | 83
  Anti-Pertussis, Booster response (N = 96, 92) | 95 | 85
  Anti-FHA, 4-Fold Increase (N = 94, 93) | 89 | 92
  Anti-FHA, Booster response (N = 94, 93) | 93 | 93

2. Primary Outcome: Geometric Mean Titers (GMTs) of Vaccine Antibodies Following Booster Vaccination With Either DTaP-Hep B-PRP~T Concomitantly With OPV or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Immunogenicity were assessed by means of enzyme immunoassay (EIA) for antibodies to the vaccine antigens 28 days after the Booster vaccination
Time Frame: Day 28 post-vaccination
Population: Geometric Mean Titers (GMTs) of Vaccine Antibodies were assessed in the per protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 98 | 98
Titers
  Anti-Hepatitis B Pre-booster (N = 98, 98) | 6.75 [5.17 to 8.81] | 17.5 [12.7 to 24.0]
  Anti-Hepatitis B Post-booster (N = 98, 98) | 119 [75.3 to 188] | 1352 [883 to 2071]
  Anti-PRP Pre-booster (N = 98, 98) | 0.908 [0.631 to 1.31] | 3.76 [2.76 to 5.13]
  Anti-PRP Post-booster (N = 98, 98) | 64.4 [47.1 to 88.2] | 103 [82.8 to 129]
  Anti-Diphtheria Pre-booster (N = 98, 98) | 0.016 [0.012 to 0.021] | 0.013 [0.010 to 0.018]
  Anti-Diphtheria Post-booster (N = 98, 98) | 2.81 [2.01 to 3.92] | 1.15 [0.779 to 1.70]
  Anti-Tetanus Pre-booster (N = 98, 98) | 0.382 [0.320 to 0.455] | 0.500 [0.429 to 0.584]
  Anti-Tetanus Post-booster (N = 98, 98) | 15.8 [13.2 to 18.9] | 14.7 [13.1 to 16.4]
  Anti-Pertussis Pre-booster (N = 96, 92) | 9.11 [7.77 to 10.7] | 6.94 [5.20 to 9.25]
  Anti-Pertussis Post-booster (N = 98, 98) | 199 [174 to 228] | 105 [76.9 to 144]
  Anti-FHA Pre-booster (N = 95, 93) | 15.0 [12.4 to 18.2] | 2.10 [1.76 to 2.51]
  Anti-FHA Post-booster (N = 97, 98) | 233 [206 to 263] | 117 [101 to 135]

3. Secondary Outcome: Number of Participants Reporting At Least 1 Solicited Injection Site and Systemic Reaction Following Booster Vaccination With Either DTaP-Hep B-PRP-T Concomitantly With Oral Polio Vaccine (OPV) or Tritanrix-Hep B/Hib™ Concomitantly With OPV
Description: Solicited injection site reactions: Tenderness, Erythema, and Swelling; Systemic reactions: Fever (Temperature), Vomiting, Crying, Somnolence, Anorexia, and Irritability.
  Grade 3 reactions are defined as: Tenderness - cries when injected limb is moved or the movement of the injected limb is reduced; Erythema and Swelling - ≥ 5cm; Fever - temperature ≥ 39.5ºC; Vomiting - ≥6 episodes per 24 hours; Crying - inconsolable crying for >3 hours; Somnolence - sleeping most of the time or difficulty to wake up; Anorexia - refuses ≥3 feeds; and Irritability - inconsolable.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Safety was assessed on the safety analysis (intent-to-treat) population.
Measure: Number; unit: Participants
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Number analyzed (Participants) | 182 | 180
Participants
  Injection site Pain | 65 | 124 [0 to 0]
  Grade 3 Injection site Pain | 1 | 9 [0 to 0]
  Injection site Erythema | 71 | 90 [0 to 0]
  Grade 3 Injection site Erythema | 2 | 1 [0 to 0]
  Injection site Swelling | 21 | 47 [0 to 0]
  Grade 3 Injection site Swelling | 1 | 2 [0 to 0]
  Extensive swelling of vaccinated limb | 0 | 0
  Pyrexia | 39 | 46 [0 to 0]
  Grade 3 Pyrexia | 0 | 2 [0 to 0]
  Vomiting | 16 | 15 [0 to 0]
  Grade 3 Vomiting | 1 | 0 [0 to 0]
  Crying | 23 | 42
  Grade 3 Crying post-vaccination | 0 | 0
  Somnolence post-vaccination | 22 | 41
  Grade 3 Somnolence | 1 | 0
  Anorexia | 24 | 39
  Grade 3 Anorexia | 1 | 0
  Irritability | 38 | 71
  Grade 3 Irritability | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to Day 28 post-vaccination.
Arm/Group | Group 1: DTaP-Hep B-PRP~T + OPV | Group 2: Tritanrix-Hep B/ Hib™ + OPV
Serious Adverse Events (participants affected / at risk) | 14/182 | 7/180
Other Adverse Events (participants affected / at risk) | 101/182 | 142/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=182) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=180)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infections (Infections and infestations) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 3 (4) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: DTaP-Hep B-PRP~T + OPV (N=182) | Group 2: Tritanrix-Hep B/ Hib™ + OPV (N=180)
Vomiting (Gastrointestinal disorders) | 16 | 15
Injection site pain (General disorders) | 65 | 124
Injection site erythemia (General disorders) | 71 | 90
Injection site swelling (General disorders) | 21 | 47
Pyrexia (General disorders) | 39 | 46
Anorexia (Metabolism and nutrition disorders) | 24 | 39
Somnolence (Nervous system disorders) | 22 | 41
Upper respiratory tract infection (Infections and infestations) | 43 | 43
Rhinitis (Metabolism and nutrition disorders) | 16 | 16
Crying (Psychiatric disorders) | 23 | 42
Irritability (Psychiatric disorders) | 38 | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications